CLINICAL TRIAL: NCT05977101
Title: A Randomized, Double-blind, Placebo-parallel Controlled Clinical Study to Evaluate the Safety and Tolerability of MY-586 SARS-CoV-2 Neutralizing Antibody Nasal Spray in Healthy Subjects
Brief Title: The Safety and Tolerability of MY-586 COVID-19 Neutralizing Antibody Nasal Spray in Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-121
Record Dates: First submitted 2022-12-27; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV-2; Prevention
Keywords: MY-586 SARS-CoV-2 Neutralizing Antibody

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MY-586 SARS-CoV-2 Neutralizing Antibody nasal spray (Experimental): Specifications: 5mg/mL, 5mL/ bottle; Provided by Chongqing Mingdao Haoyue Biotechnology Co., LTD
  Interventions: Biological: MY-586 SARS-CoV-2 Neutralizing Antibody nasal spray
- MY-586 SARS-CoV-2 Neutralization Antibody nasal excipient (Placebo Comparator): Specifications: 0mg/mL, 5mL/ bottle; Provided by Chongqing Mingdao Haoyue Biotechnology Co., LTD
  Interventions: Other: Placebo Comparator: MY-586 SARS-CoV-2 Neutralization Antibody nasal excipient

INTERVENTIONS:
Biological: MY-586 SARS-CoV-2 Neutralizing Antibody nasal spray — Patients who met the inclusion and exclusion criteria were randomly assigned to one of three different cohorts. Subjects in each cohort were randomly assigned in a ratio of 5:1 to two parallel dosing groups, one of which served as the control group. Each cohort was given either an experimental drug or a placebo nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose, and left nasal swabs and throat swabs were collected for immunotoxicity and drug concentration testing.
  Arms: MY-586 SARS-CoV-2 Neutralizing Antibody nasal spray
Other: Placebo Comparator: MY-586 SARS-CoV-2 Neutralization Antibody nasal excipient — Patients who met the inclusion and exclusion criteria were randomly assigned to one of three different cohorts. Subjects in each cohort were randomly assigned in a ratio of 5:1 to two parallel dosing groups, one of which served as the control group. Each cohort was given either an experimental drug or a placebo nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose, and left nasal swabs and throat swabs were collected for immunotoxicity and drug concentration testing.
  Arms: MY-586 SARS-CoV-2 Neutralization Antibody nasal excipient

SUMMARY:
This is a randomized, double-blind, placebo-parallel intervention clinical study that will include approximately 72 healthy subjects based on inclusion and exclusion criteria. Patients who met the inclusion and exclusion criteria were randomly assigned to one of three different cohorts. Subjects in each cohort were randomly assigned in a ratio of 5:1 to two parallel dosing groups, one of which served as the control group. Each cohort was given either an experimental drug or a placebo nasal spray at different doses and intervals, and blood was collected on an empty stomach before the first dose, and left nasal swabs and throat swabs were collected for immunotoxicity and drug concentration testing. 14 days after the last dose, subjects will return to the study Center for blood samples, left nasal swabs, and throat swabs to be collected for drug concentration, immunotoxicity, and safety laboratory indicators (routine blood and biochemistry). To evaluate the safety and tolerability of MY-586 SARS-CoV-2 Neutralizing Antibody nasal spray in healthy subjects, and to evaluate its serum concentrations and nasal and pharyngeal swab concentrations by comparing the test results of different cotillaries.

DETAILED DESCRIPTION:
As of December 5, 2021, more than 266 million COVID-19 cases and 5.26 million deaths have been reported worldwide, according to Worldometer Real-time statistics. On 27 November 2021, a highly mutated new variant of COVID-19 (named Omicron by the WHO) was discovered in South Africa. Although the introduction of vaccines has played a huge role in the prevention and control of COVID-19, the neutralizing antibodies stimulated by different vaccines differ greatly, and the antibody maintains a high titer in the human body for a short time (3-6 months at most), so the global demand for safe and effective prevention of COVID-19 remains unmet.

The novel coronavirus neutralizing antibody can directly bind to the envelope of the novel coronavirus to rapidly block the virus infection, which has been fully verified as a safe and effective treatment. But so far, there are no approved antibodies at home or abroad to prevent infection with the novel coronavirus, In addition, there is a lack of broad-spectrum monoclonal neutralizing antibodies with high efficiency against mutant strains (currently, all the approved neutralizing antibodies in the world are used in combination with two antibodies), which can be used as reference for the administration of neutralizing antibodies for the prevention of a wide range of people (intravenous infusion as the prophylactic administration will lead to low compliance of the administration population).

MY-586, a SARS-CoV-2 Neutralizing Antibody, was screened from peripheral blood lymphocytes of patients recovering from COVID-19, and 209 strains of SARS-CoV-2-specific antibody were isolated from them, among which MY-586 was a super antibody with strong and effective neutralizing effect on the novel coronavirus and the circulating strains of UK, India, South Africa and India Delta.

Currently, the evaluation of the preclinical efficacy and safety of MY-586 SARS-CoV-2 Neutralizing Antibody and the production of CMC to support clinical trials are nearing completion. All the data showed that MY-586 SARS-CoV-2 Neutralizing Antibody had excellent efficacy, safety and druggability. In particular, MY-586 SARS-CoV-2 Neutralizing Antibody is administered by nasal spray. Although there are no approved nasal spray neutralizing antibody drugs on the market at home and abroad, the investigators have successfully solved the drugging of MY-586 SARS-CoV-2 Neutralizing Antibody by nasal spray and the development of nasal spray device. The nasal spray type MY-586 SARS-CoV-2 Neutralizing Antibody is easy to carry, easy to administer, and has strong accessibility and compliance for the population. It can be used as a new and widely used safe and effective preventive measure besides vaccines. Therefore, the rapid clinical research and development of MY-586 SARS-CoV-2 Neutralizing Antibody will provide a more effective guarantee for social safety and effective prevention of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand the purpose, nature, method and possible adverse reactions of the experiment, voluntarily participate in the experiment, and sign informed consent before the experiment begins;
2. Healthy subjects aged 18-65 years (including the critical value) with an appropriate sex ratio between men and women;
3. Body Mass index (BMI) = weight (kg)/height 2 (m2), with a BMI in the range of 19.0 to 30.0 (including the cutoff). Male subjects should weigh at least 50.0kg and female subjects should weigh at least 45.0kg;
4. The subjects had no birth plan for 3 months from the date of signing the informed consent to the end of the study, and agreed to voluntarily take effective and appropriate contraceptive measures with their partners during this period;
5. Negative nucleic acid test of novel coronavirus;
6. Subjects can communicate well with researchers and understand and comply with the requirements of this study.

Exclusion Criteria:

1. Allergic to any ingredient in this product and auxiliary materials; Or allergic (such as allergic to two or more drugs, food);
2. Patients with symptoms of acute upper respiratory tract infection within 1 week before administration;
3. Patients with acute episodes of chronic rhinitis or anatomical abnormalities affecting drug absorption in the nose;
4. Patients with a history of asthma;
5. Asplenia or functional asplenia caused by any condition;
6. Diseases or factors with clinical abnormalities that need to be excluded, including but not limited to diseases of the nervous system, cardiovascular system, kidney, liver, gastrointestinal system, respiratory system, metabolism, bone system and other systems;
7. Vital signs, physical examination, laboratory examination (such as white blood cell count less than 3.0*109/L, platelet count less than 75*109/L, TB > 1.5*ULN, ALT > 1*ULN, AST > 1*ULN) and electrocardiogram examination of any items abnormal and judged by the investigator to be clinically significant;
8. Use of any prescription or over-the-counter drugs within 14 days before administration;
9. Patients who had received immunosuppressive therapy, cytotoxic therapy or inhaled corticosteroid therapy within 6 months before administration;
10. A history of drug abuse or use of any drug in the 6 months prior to drug administration;
11. Pregnant and lactating women;
12. The subject has not taken effective and appropriate contraceptive measures within 30 days before the drug administration;
13. The subjects had sperm and egg donation plans within 3 months after the first drug administration to the end of the study;
14. Blood donation or massive blood loss (≥200mL), receiving blood transfusion or using blood products within 3 months prior to drug administration; Or plan to donate blood or blood components during the trial;
15. Have participated in other drug clinical trials or device clinical trials, and have taken test drugs or used test devices within 3 months before drug administration;
16. Subjects may not be able to comply with the protocol to complete the study for other reasons or the investigator may decide that it is not suitable for participants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
vital signs | 14 days before the trial,1 days before the trial, after each dose
  Including pulse, blood pressure, temperature
laboratory tests | Including blood routine, blood biochemistry, routine urine pregnancy test (female) limited
  Including blood routine, blood biochemistry, routine urine pregnancy test (female) limited
12-lead electrocardiogram | 14 days before the trial,1 days before the trial, after each dose
  Including ECG QT Interval、PR Interval
adverse events | Up to 1 year
  Adverse reactions were recorded by questionnaire. Observe any adverse events

SECONDARY OUTCOMES:
Drug concentration index | 15 minutes after each dose
  Drug concentration of serum, nasal swab and pharyngeal swab
Immunotoxicity detection indicators | 15 minutes after each dose
  Serum autoantibody titer
Cytokines | 15 minutes after each dose
  Serum Cytokines titer
lymphocyte subsets | 15 minutes after each dose
  Serum lymphocyte subsets

CONTACTS AND LOCATIONS:
Overall Officials: Dazhi Zhang, M.D., Study Chair — The Second Affiliated Hospital of Chongqing Medical University
Locations (1):
- The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No